CLINICAL TRIAL: NCT03375489
Title: Comparative Effectiveness of Early Integrated Telehealth Versus In-Person Palliative Care for Patients With Advanced Lung Cancer
Brief Title: Early Integrated Telehealth Versus In-Person Palliative Care for Patients With Lung Cancer
Acronym: REACH PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Palliative Care Research Cooperative Group (Network)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-484; R-1609-35995 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute)
Record Dates: First submitted 2017-11-30; First posted 2017-12-18 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer palliative care
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Palliative Care (Experimental): * Patient and caregiver will meet with the palliative care clinician in person within four weeks of enrollment.
  * Subsequent visits with the palliative care clinician will be conducted with the patient and caregiver in their home or other location using video at least every four weeks.
  * Patient and caregiver may be scheduled to meet with the palliative care clinician in the clinic if requested by the patient or a clinician.
  (Note: Caregiver enrollment in the study and attendance at palliative care visits are voluntary, and the patient can participate with no enrolled caregiver.)
  Interventions: Other: Telehealth Palliative Care
- In-person Palliative Care (Active Comparator): * Patient and caregiver will be scheduled for their first in-person palliative care visit within four weeks of enrollment and then at least every four weeks thereafter until the patient is no longer coming into the clinic.
  * In-person palliative care visits will be scheduled on the same day as an oncology visit if possible.
  (Note: Caregiver enrollment in the study and attendance at palliative care visits are voluntary, and the patient can participate with no enrolled caregiver.)
  Interventions: Other: In-person Palliative Care

INTERVENTIONS:
Other: Telehealth Palliative Care — Teleconference meeting with the palliative care team. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
  Arms: Telehealth Palliative Care
Other: In-person Palliative Care — In-person meeting with the palliative care team. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
  Arms: In-person Palliative Care

SUMMARY:
This research study is evaluating ways to provide palliative care to patients who have recently been diagnosed with lung cancer and their families.

DETAILED DESCRIPTION:
Patients with serious cancers, like advanced lung cancer, often experience physical symptoms, such as pain or shortness of breath. In addition, both patients and their loved ones (family and friends) often feel worried or sad about the cancer diagnosis.

Research has shown that early involvement of a team of clinicians that specialize in lessening (or "palliating") many of these distressing physical and emotional symptoms and in helping patients and their families cope with a serious illness improves patients' and their loved ones' experience with their cancer. This team is called "palliative care," and consists of physicians and advanced practice nurses (or "nurse practitioners") who work closely and collaboratively with the oncology team to care for the participant and the participant's loved ones. Research shows that when the palliative care team works closely with the oncology team to care for patients with advanced cancer, they have better symptom control, quality of life, and mood, and their loved ones feel less distressed. the investigators call this model of care, "early integrated palliative care."

While the investigators know that having palliative care clinicians work closely with the oncology team is helpful for patients and their loved ones, many patients do not have access to these specialists because hospitals and cancer clinics lack enough staff and because some patients and family members live in distant regions that make attending clinic visits difficult and expensive. One way to overcome these barriers is to have patients meet with palliative care clinicians using secure video-conferencing technology.

The purpose of this study is to determine if meeting with a palliative care clinician through video-conferencing is just as beneficial for patients and their families as meeting with a palliative care clinician in person. Specifically, this study will compare these two different strategies for meeting with the palliative care clinician. The first strategy is to schedule the participant to meet with the palliative care clinician regularly each month in person at the clinic. The investigators call this strategy "In-person palliative care."

The second strategy is to schedule the participant to meet with the palliative care clinician regularly each month using secure video-conferencing, such as through a smart phone or tablet computer. If the participant do not have this form of technology, the investigators will provide it for the participant. The investigators call this strategy "telehealth palliative care." The primary goals of this study are to learn if telehealth palliative care is just as effective as in-person palliative care for improving quality of life, mood symptoms, and satisfaction with care for patients with advanced lung cancer and their families.

ELIGIBILITY:
Inclusion Criteria:

* Patient Eligibility Criteria

  * Diagnosed with advanced non-small cell lung cancer being treated with non-curative intent, and informed of advanced disease within the prior twelve weeks
  * Eastern Cooperative Oncology Group (ECOG) Performance Status from 0 (asymptomatic) to 3 (symptomatic and in bed >50% of the day)
  * The ability to read and respond to questions in English or Spanish
  * Receiving primary cancer care at one of the participating sites
  * Age > or = 18 years
  * Lives in a state where their institutions' palliative care clinicians are licensed to practice
* Caregiver Eligibility Criteria

  * Relative or friend who is identified by the patient participant and lives with the patient or has contact with them at least twice per week
  * The ability to read and respond to questions in English or Spanish
  * Age > or = 18 years

Exclusion Criteria:

* Patient Exclusion Criteria

  * Already receiving outpatient palliative care or hospice services
  * Cognitive or psychiatric conditions as determined by the treating oncologist to prohibit study consent or participation
* Caregiver Exclusion Criteria

  * Cognitive or psychiatric conditions as determined by the treating oncologist to prohibit study consent or participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1798 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (23):
- United States (23):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Los Angeles, California
  - University of California - San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Dartmouth-Hitchcock Health, Lebanon, New Hampshire
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas at Austin, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Greer JA, Temel JS, El-Jawahri A, Rinaldi S, Kamdar M, Park ER, Horick NK, Pintro K, Rabideau DJ, Schwamm L, Feliciano J, Chua I, Leventakos K, Fischer SM, Campbell TC, Rabow MW, Zachariah F, Hanson LC, Martin SF, Silveira M, Shoemaker L, Bakitas M, Bauman J, Spoozak L, Grey C, Blackhall L, Curseen K, O'Mahony S, Smith MM, Rhodes R, Cullinan A, Jackson V; REACH PC Investigators. Telehealth vs In-Person Early Palliative Care for Patients With Advanced Lung Cancer: A Multisite Randomized Clinical Trial. JAMA. 2024 Sep 11;332(14):1153-64. doi: 10.1001/jama.2024.13964. Online ahead of print. PMID 39259563
- [Derived] Petrillo LA, El-Jawahri A, Heuer LB, Post K, Gallagher ER, Trotter C, Elyze M, Vyas C, Plotke R, Turk YR, Han J, Temel JS, Greer JA. Health-Related Quality of Life and Depression Symptoms in a Cross Section of Patients with Advanced Lung Cancer before and during the COVID-19 Pandemic. J Palliat Med. 2022 Nov;25(11):1639-1645. doi: 10.1089/jpm.2022.0049. Epub 2022 May 19. PMID 35588200

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Note: Caregiver enrollment in the study and attendance at palliative care visits were voluntary, and patients could participate without an enrolled caregiver. Only one caregiver per patient participant was invited to enroll in the study.
Groups:
- Telehealth Palliative Care: Patient: * Patient and caregiver will meet with the palliative care clinician in person within four weeks of enrollment.
  * Subsequent visits with the palliative care clinician will be conducted with the patient and caregiver in their home or other location using video at least every four weeks.
  * Patient and caregiver may be scheduled to meet with the palliative care clinician in the clinic if requested by the patient or a clinician.
  Telehealth Palliative Care: Teleconference meeting via video with the palliative care team. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
- In-person Palliative Care: Patient; In-person Palliative Care: Caregiver: * Patient and caregiver will be scheduled for their first in-person palliative care visit within four weeks of enrollment and then at least every four weeks thereafter until the patient is no longer coming into the clinic.
  * Palliative care visits will be scheduled on the same day as an oncology visit if possible.
  In-person Palliative Care: In-person meeting with the palliative care team in clinic. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
- Telehealth Palliative Care: Caregiver: * Patient and caregiver will meet with the palliative care clinician in person within four weeks of enrollment.
  * Subsequent visits with the palliative care clinician will be conducted with the patient and caregiver in their home or other location using video at least every four weeks.
  * Patient and caregiver may be scheduled to meet with the palliative care clinician in the clinic if requested by the patient or a clinician.
Period: Overall Study
Arm/Group | Telehealth Palliative Care: Patient | In-person Palliative Care: Patient | Telehealth Palliative Care: Caregiver | In-person Palliative Care: Caregiver
Started | 633 (Number represents total patients enrolled and assigned to the Telehealth Palliative Care Group.) | 617 (Number represents total patients enrolled and assigned to the In-person Palliative Care Group.) | 272 (Number represents total caregivers enrolled and assigned to the Telehealth Palliative Care Group in tandem with the respective patient participant.) | 276 (Number represents total caregivers enrolled and assigned to the In-person Palliative Care Group in tandem with the respective patient participant.)
Completed | 633 | 617 | 272 | 276
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population represents the 1250 patients enrolled in the study (i.e., 633 patients assigned to the Telehealth Palliative Care Group and 617 patients assigned to the In-person Palliative Care Group) as well as the 548 caregivers enrolled in the study (i.e., 272 caregivers assigned to the Telehealth Palliative Care Group and 276 caregivers assigned to the In-person Palliative Care Group in tandem with the respective patient participant).
Groups:
- Telehealth Palliative Care: Patient; Telehealth Palliative Care: Caregiver: * Patient and caregiver will meet with the palliative care clinician in person within four weeks of enrollment.
  * Subsequent visits with the palliative care clinician will be conducted with the patient and caregiver in their home or other location using video at least every four weeks.
  * Patient and caregiver may be scheduled to meet with the palliative care clinician in the clinic if requested by the patient or a clinician.
  (Note: Caregiver enrollment in the study and attendance at palliative care visits are voluntary, and the patient can participate without an enrolled caregiver.)
  Telehealth Palliative Care: Teleconference meeting via video with the palliative care team. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
- In-person Palliative Care: Patient; In-person Palliative Care: Caregiver: * Patient and caregiver will be scheduled for their first in-person palliative care visit within four weeks of enrollment and then at least every four weeks thereafter until the patient is no longer coming into the clinic.
  * In-person palliative care visits will be scheduled on the same day as an oncology visit if possible.
  (Note: Caregiver enrollment in the study and attendance at palliative care visits are voluntary, and the patient can participate without an enrolled caregiver.)
  In-person Palliative Care: In-person meeting with the palliative care team in clinic. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
- Total: Total of all reporting groups
Arm/Group | Telehealth Palliative Care: Patient | In-person Palliative Care: Patient | Telehealth Palliative Care: Caregiver | In-person Palliative Care: Caregiver | Total
Number analyzed (Participants) | 633 | 617 | 272 | 276 | 1798
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Four caregiver participants in the Telehealth Palliative Care Group and two caregiver participants in the In-person Palliative Care group did not complete the age question on the socio-demographic questionnaire, and therefore their baseline age data are missing.
  years
    number analyzed (Participants) | 633 | 617 | 268 | 274 | 1792
    (all) | 65.5 (10.9) | 65.5 (10.6) | 56.8 (14.8) | 58.0 (13.2) | 63.0 (12.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 356 | 318 | 182 | 194 | 1050
  Man | 277 | 297 | 90 | 82 | 746
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 30 | 10 | 14 | 83
  Not Hispanic or Latino | 596 | 575 | 255 | 255 | 1681
  Unknown or Not Reported | 8 | 12 | 7 | 7 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was collected by self-report, which allowed multiple selections from a predetermined list, including an "other" (write-in) option. Sum of percentages may exceed 100%. In the Telehealth Palliative Care Group, 21 patients and 7 caregivers self-identified as an "other" racial category that was not provided as an option. In the In-person Palliative Care Group, 10 patients and 2 caregivers self-identified as an "other" racial category that was not provided as an option.
  Participants
    American Indian or Alaska Native | 4 | 4 | 2 | 1 | 11
    Asian | 32 | 32 | 9 | 12 | 85
    Black or African American | 57 | 72 | 17 | 22 | 168
    Native Hawaiian or Other Pacific Islander | 2 | 4 | 0 | 2 | 8
    White | 524 | 502 | 238 | 235 | 1499
    Other | 21 | 10 | 7 | 2 | 40
    Unknown or Not Reported | 3 | 6 | 1 | 4 | 14
Region of Enrollment [Number; unit: participants]
  United States | 633 | 617 | 272 | 276 | 1798

OUTCOME MEASURES:

1. Primary Outcome: Patient-reported Quality of Life
Description: Compare the difference between study groups in patient-reported quality of life as measured by the Functional Assessment of Cancer Therapy - Lung Questionnaire, which has a total scale score range from 0-136 with higher scores indicating better overall quality of life.
Time Frame: 24 Weeks
Population: The analysis population represents the numbers of patients in each study group who completed the baseline and 24-week Functional Assessment of Cancer Therapy - Lung Questionnaire.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Telehealth Palliative Care: Patients: * Patient and caregiver will meet with the palliative care clinician in person within four weeks of enrollment.
  * Subsequent visits with the palliative care clinician will be conducted with the patient and caregiver in their home or other location using video at least every four weeks.
  * Patient and caregiver may be scheduled to meet with the palliative care clinician in the clinic if requested by the patient or a clinician.
  (Note: Caregiver enrollment in the study and attendance at palliative care visits are voluntary, and the patient can participate without an enrolled caregiver.)
  Telehealth Palliative Care: Teleconference meeting via video with the palliative care team. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
- In-person Palliative Care: Patients: * Patient and caregiver will be scheduled for their first in-person palliative care visit within four weeks of enrollment and then at least every four weeks thereafter until the patient is no longer coming into the clinic.
  * In-person palliative care visits will be scheduled on the same day as an oncology visit if possible.
  (Note: Caregiver enrollment in the study and attendance at palliative care visits are voluntary, and the patient can participate without an enrolled caregiver.)
  In-person Palliative Care: In-person meeting with the palliative care team in clinic. Palliative care is a medical specialty focused on lessening (or "palliating") patients' symptoms and helping patients and their families cope with a serious illness.
Arm/Group | Telehealth Palliative Care: Patients | In-person Palliative Care: Patients
Number analyzed (Participants) | 305 | 315
units on a scale | 99.7 [98.0 to 101.3] | 97.7 [96.1 to 99.3]
Statistical Analysis 1: Comparison: Telehealth Palliative Care: Patients vs In-person Palliative Care: Patients; The difference in week-24 means between groups was estimated using a linear regression model with a main effect for group assignment and controlling for baseline Functional Assessment of Cancer Therapy - Lung Questionnaire scores; Test type: Equivalence — Equivalence was established for patient-reported quality of life if the 90% confidence interval for the estimated difference in means was within the margin of ±4 points on the Functional Assessment of Cancer Therapy - Lung Questionnaire; p = 0.04, Regression, Linear — The a priori threshold for statistical significance was p<0.05; Mean Difference (Final Values) = 2.0, 90% CI 2-sided [0.1 to 3.9]

2. Secondary Outcome: Patient-reported Communication About Their End-of-Life Care Preferences With Their Clinicians
Description: Compare the difference between study groups in the proportion of patients who reported that they discussed their end-of-life care preferences with their clinicians based on a single item from the Prognosis and Treatment Perceptions Questionnaire (PTPQ). The PTPQ includes a self-report item that assesses whether the patient communicated with their clinicians about their wishes for care if they were dying (i.e., scored dichotomously as "yes vs. no").
Time Frame: 48 weeks (or last assessment prior to death if before 48 weeks)
Population: The analysis population represents the numbers of patients in each study group who completed the Prognosis and Treatment Perceptions Questionnaire at least once post baseline up to 48 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Telehealth Palliative Care: Patients | In-person Palliative Care: Patients
Number analyzed (Participants) | 446 | 442
Participants | 130 | 115
Statistical Analysis 1: Comparison: Telehealth Palliative Care: Patients vs In-person Palliative Care: Patients; The difference between groups in the proportions of patients reporting that they communicated with their clinicians about their end-of-life care preferences was estimated using a binomial generalized estimating equation model with robust standard errors, the identity link function, and a main effect for group assignment; Test type: Equivalence — Equivalence was established for patient-reported communication with their clinicians about their end-of-life care preferences if the 90% confidence interval for the estimated difference in proportions was within the margin of ±8%; p = 0.26, binomial generalized estimating equation — Bonferroni-adjusted p-value; Estimated Difference in Proportions = 3.1, 90% CI 2-sided [-1.8 to 8.1]

3. Secondary Outcome: Length of Stay in Hospice
Description: Compare the difference between study groups in the length of stay in hospice (as measured in days) among patients who died during study period per medical record review.
Time Frame: From hospice enrollment until patient death during study period
Population: The analysis population represents the numbers of patients in each study group who who died during the study period.
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Telehealth Palliative Care: Patients | In-person Palliative Care: Patients
Number analyzed (Participants) | 360 | 363
days | 25.3 [19.2 to 31.3] | 25.1 [19.0 to 31.1]
Statistical Analysis 1: Comparison: Telehealth Palliative Care: Patients vs In-person Palliative Care: Patients; The difference in mean length of stay in hospice between groups was estimated using a linear regression model with a main effect for group assignment; Test type: Equivalence — Equivalence was established for patient length of stay in hospice if the 90% confidence interval for the estimated difference in mean days was within the margin of ±6 days; p = 0.46, Regression, Linear — Bonferroni-adjusted p-value; Mean Difference (Final Values) = 0.2, 90% CI 2-sided [-7.0 to 7.4]

4. Secondary Outcome: Proportion of Patient's Palliative Care Visits With a Caregiver Present
Description: Compare the difference between study groups in the proportion of palliative care visits that had a caregiver present as documented by the palliative care clinician using a study visit summary form.
Time Frame: 24 weeks
Population: The analysis population represents the numbers of patients in each study group who had any palliative care visits, and the overall number of units analyzed represents the numbers of palliative care visits in each study group through week 24.
Measure: Number (95% Confidence Interval); unit: proportion of visits with a caregiver
Units Other Than Participants: Number of Palliative Care Visits
Arm/Group | Telehealth Palliative Care: Patient | In-person Palliative Care: Patient
Number analyzed (Participants) | 576 | 549
Number analyzed (Number of Palliative Care Visits) | 2618 | 2588
proportion of visits with a caregiver | 36.6 [33.6 to 39.7] | 49.7 [46.4 to 53.1]
Statistical Analysis 1: Comparison: Telehealth Palliative Care: Patient vs In-person Palliative Care: Patient; The proportion of palliative care visits with caregiver participation was compared using a binomial generalized estimating equation model with robust standard errors, the identity link function, and a main effect for group assignment; Test type: Superiority; p < 0.001, binomial generalized estimating equation — Bonferroni-adjusted p-value; Difference in estimated proportions = -13.0, 95% CI 2-sided [-17.6 to -8.6]

5. Secondary Outcome: Patient-reported Satisfaction With Care
Description: Compare the difference between study groups in patient-reported satisfaction with care as measured by the Satisfaction and Care Delivery Questionnaire, which has a total scale score range from 0-52 with higher scores indicating greater satisfaction.
Time Frame: 24 weeks
Population: The analysis population represents the numbers of patients in each study group who completed the 24-week Satisfaction and Care Delivery Questionnaire.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Telehealth Palliative Care: Patient | In-person Palliative Care: Patient
Number analyzed (Participants) | 422 | 422
units on a scale | 41.3 [40.4 to 42.3] | 41.0 [40.1 to 41.9]
Statistical Analysis 1: Comparison: Telehealth Palliative Care: Patient vs In-person Palliative Care: Patient; The difference in week-24 means between groups was estimated using a linear regression model with a main effect for group assignment; Test type: Superiority; p > 0.99, Regression, Linear — Bonferroni-adjusted p-value; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-1.0 to 1.7]

6. Secondary Outcome: Caregiver-reported Satisfaction With Care
Description: Compare the difference between study groups in caregiver-reported satisfaction with care as measured by the Satisfaction and Care Delivery Questionnaire (caregiver version), which has a total scale score range from 0-48 with higher scores indicating greater satisfaction.
Time Frame: 24 weeks
Population: The analysis population represents the numbers of caregivers in each study group who completed the 24-week Satisfaction and Care Delivery Questionnaire.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Telehealth Palliative Care: Caregiver | In-person Palliative Care: Caregiver
Number analyzed (Participants) | 176 | 177
units on a scale | 37.2 [35.8 to 38.5] | 36.8 [35.4 to 38.2]
Statistical Analysis 1: Comparison: Telehealth Palliative Care: Caregiver vs In-person Palliative Care: Caregiver; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p > 0.99, Regression, Linear — Bonferroni-adjusted p-value; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.5 to 2.3]

7. Other Pre Specified Outcome: Patient-reported Coping Strategies
Description: Compare the difference between study groups in patient-reported coping strategies as measured by the Brief Cope (approach-oriented coping score range: 6-24, with higher scores indicating greater use of approach-oriented coping strategies; avoidant coping score range: 4-16, with higher scores indicating greater use of avoidant coping strategies).
Time Frame: up to 48 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Patient-reported Prognostic Understanding
Description: Compare the difference between study groups in patient-reported prognostic understanding as measured by the Prognosis and Treatment Perceptions Questionnaire, in which patients rate two items about the goal of their cancer care (i.e., scored dichotomously as either "to cure my cancer" vs any other option) and whether their cancer is curable (i.e., scored dichotomously as "yes or no").
Time Frame: up to 48 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Caregiver-reported Prognostic Understanding
Description: Compare the difference between study groups in caregiver-reported prognostic understanding as measured by the Prognosis and Treatment Perceptions Questionnaire, in which caregivers rate two items about the goal of their loved one's cancer care (i.e., scored dichotomously as either "to cure his/her cancer" vs any other option) and whether their loved one's cancer is curable (i.e., scored dichotomously as "yes or no").
Time Frame: up to 48 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Caregiver-reported Quality of Life
Description: Compare the difference between study groups in caregiver-reported quality of life as measured by the Caregiver Oncology Quality of Life Questionnaire, which has a total scale score range of 0-100 with higher scores indicating better quality of life.
Time Frame: up to 48 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Caregiver-reported Mood Symptoms
Description: Compare the difference between study groups in caregiver-reported mood symptoms as measured by the Hospital Anxiety and Depression Scale (anxiety subscale score range, 0-21, with higher scores indicating greater anxiety symptoms; depression subscale score range, 0-21, with higher scores indicating greater depression symptoms).
Time Frame: up to 48 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Patient-reported Mood Symptoms
Description: Compare the difference between study groups in patient-reported mood symptoms as measured by the Hospital Anxiety and Depression Scale (anxiety subscale score range, 0-21, with higher scores indicating greater anxiety symptoms; depression subscale score range, 0-21, with higher scores indicating greater depression symptoms).
Time Frame: up to 48 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Patient-reported Depression
Description: Compare the difference between study groups in patient-reported depression as measured by the Patient Health Questionnaire-9, which has a total scale score range from 0-27 with higher scores indicating more significant depression symptoms.
Time Frame: up to 48 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Health Care Utilization
Description: Compare the difference between study groups in health care utilization as per medical record review of emergency department visits, hospital admissions, chemotherapy administration at the end of life, and hospice service use.
Time Frame: Through study completion, average of 18 month follow up
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Caregiver-reported Quality of Patient Death
Description: Compare the difference between study groups in caregiver-reported quality of patient death as measured by the After Death Assessment, which includes three items that ask the caregiver to rate the quality of the patient's death (from 1 "worst possible" to 10 "best possible"), the degree of physical distress the patient experienced in their last week of life (from 1 "none" to 10 "extremely distressed"), and the degree of psychological distress the patient experienced in their last week of life (from 1 "none" to 10 "extremely upset").
Time Frame: Up to 6 months after patient death during study period
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Patient-reported Quality of Life
Description: Compare the difference between study groups in patient-reported quality of life across all study assessment time points as measured by the Functional Assessment of Cancer Therapy - Lung Questionnaire, which has a total scale score range from 0-136 with higher scores indicating better quality of life.
Time Frame: up to 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 18 months post enrollment.
Description: No serious or other (non-serious) adverse events were collected or monitored in this minimal risk supportive care trial for patient or caregiver participants. As a result, the total number of patient and caregiver participants at risk for adverse events is zero since this was not monitored in this supportive care trial. Mortality data for caregiver participants were not collected as part of this study.
Arm/Group | Telehealth Palliative Care: Patients | In-person Palliative Care: Patients
All-Cause Mortality (participants affected / at risk) | 365/633 | 368/617
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT03375489/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03375489/SAP_001.pdf